CLINICAL TRIAL: NCT03180424
Title: Impact on Functional Status in Older Adults Treated With L-Carnitine
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Clínicas Dr. Manuel Quintela (Other)
Collaborators: University of the Republic, Uruguay (Other)
Responsible Party: Principal Investigator, Ana Barboza, Principal Investigator, Hospital de Clínicas Dr. Manuel Quintela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocolo L-Carnitina
Record Dates: First submitted 2017-05-31; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Carnitine; Muscle; Functional Status; Old Age; Debility
Keywords: carnitine; elderly; functional status
MeSH Terms: conditions — Frailty | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- L Carnitine + Exercise at home (Active Comparator): Patients who will receive L Carnitine, in liquid form, at a dosage of 2g per day, in a single intake, in addition to physical exercise advice at home for which a manual will be delivered in the consultation, for 12 weeks.
  Interventions: Drug: L Carnitine; Behavioral: Exercise at home
- L Carnitine + supervised exercise (Experimental): Patients receiving L Carnitine, in liquid form, at doses of 2g per day, in a single intake, in addition to a supervised physical exercise plan, for 12 weeks.
  Interventions: Drug: L Carnitine; Behavioral: Supervised exercise
- Placebos + supervised exercise (Placebo Comparator): Patients receiving placebo and supervised exercise plan.
  Interventions: Behavioral: Supervised exercise; Drug: Placebos

INTERVENTIONS:
Drug: L Carnitine — L Carnitine liquid, single daily dose of 2g orally.
  Arms: L Carnitine + Exercise at home; L Carnitine + supervised exercise
Behavioral: Supervised exercise — Modified Otago exercise programme, 2 times a week with a duration of 45 minutes, to be supervised by a previously qualified and trained instructor. Follow up of the established plan includes an adequate monitoring, evaluating the evolution and the possible adverse effects that may appear.
  Arms: L Carnitine + supervised exercise; Placebos + supervised exercise
Drug: Placebos — Liquid substance, similar to the one containing L carnitine, in the same presentation
  Arms: Placebos + supervised exercise
Behavioral: Exercise at home — A schedule of exercises will be given in the consultation, which the patient will perform at home, without supervision
  Arms: L Carnitine + Exercise at home

SUMMARY:
This study evaluates the impact of the treatment with L-Carnitine on the function of adults over 65 years, in conjunction with regular exercise. Simple randomization will be performed, distributing patients in 3 treatment groups, with L-Carnitine or Placebo, and with physical exercise at home or supervised.

DETAILED DESCRIPTION:
The supplemental intake of L-carnitine improves the physical functioning of the pre-fragile and fragile elder of the community.

Circulating L-carnitine levels increase after administration of the supplement. The impact on the function of L-carnitine in combination with physical exercise will be studied in a population of older adults in Montevideo.

The sample will be divided into 3 groups, according to the intervention:

Group 1: Patients who will receive L-Carnitine in addition to a manual to perform physical exercise at home.

Group 2: Patients receiving L-Carnitine plus supervised exercise plan. Group 3: Patients receiving placebo and supervised exercise plan. All three groups will be evaluated for functional and anthropometric parameters: prior, during and after intervention. In addition, the dosage of L-carnitine and acetylcarnitine will be evaluated before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet at least 2 criteria for the fragility phenotype of Linda Fried
* Ability to comply with aerobic physical activity of moderate intensity and basic resistance.
* Not depressed patients (Yesavage <5 in patients without previous depression or Hamilton <7 in patients in treatment for depression)
* MMSE (Mini-Mental State Examination) greater than 24 points.
* Independent or mildly dependent patients, Barthel> 95 points.
* Patients without visual disturbances or with decreased visual acuity corrected.
* No pain or with VAS (Visual analogue scale) <3/10.
* Patients without nutritional risk, MNA (Mini Nutritional Assessment > 23.5 / 30 points) and BMI (Body Mass Index) > 23 kg / m2.

Exclusion Criteria:

* Absolute contraindications for performing physical exercise: recent AMI or unstable angina, uncontrolled hypertension, acute HF and complete AV block.
* Patients with osteoarticular pathology that limits their physical activity.
* Previous neurological pathology (Stroke, Enf. Of Parkinson's).
* Acute or chronic diseases decompensated or with lymphedema that makes difficult the accomplishment of the bioimpedanciometry.
* Patients using orthopedic devices and prostheses or pacemakers that interfere with gait or impede the achievement of bioimpedanciometry.
* BMI less than 23 and / or an involuntary weight loss of 3kg or more in the last 3 months.
* Psychiatric disorders that hinder adherence to treatment.
* Moderate to severe Chronic Renal Disease
* Patient who does not agree to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-08-31 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in elderly's function | 12 weeks
  Independence Scales for Activities of Daily Living
Gait speed | 12 weeks
  Gait speed measured after the intervention
Elderly's physical performance | 12 weeks
  Elderly's physical performance assessed by SPPB (Short Physical Performance Battery Protocol).

SECONDARY OUTCOMES:
Changes in the expression of fragility criteria | 12 weeks
  The Fragility criteria will be measured according to criteria promulgated and validated by Fried. The 5 original criteria will be used, but some measures to characterize the fragility will be adapted to the modifications of Avila-Funes.

OTHER OUTCOMES:
Determine blood levels of L carnitine and acetylcarnitine | 12 weeks
  Determine L-Carnitine and Acetylcarnitine levels in the study population before and after L carnitine supplementation.
Determine levels of ammonia in blood | 12 weeks
  Determine levels of ammonia in blood in the study population before and after L carnitine supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Sgaravatti, MD, Study Director — HospítalCDMQ
Locations (1):
- Hospital de Clinicas Dr. Manuel Quintela, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: Undecided